CLINICAL TRIAL: NCT02311790
Title: Supplementation With Vegetable Oils Enriched in the Fatty Acids Trans-C16:1 or Cis-C16:1: Dose-response Study
Brief Title: Palmitoleic Isomer Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 11516
Record Dates: First submitted 2014-12-04; First posted 2014-12-08 (Estimated); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Insulin Sensitivity
Keywords: cis-C16:1n7 supplement; trans-C16:1n7 supplement; palmitoleic acid supplement
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Trans-C16:1 supplement (Experimental): Volunteers will take trans-C16:1 supplement for 3 weeks
  Interventions: Dietary Supplement: Trans-C16:1 supplement
- Cis-C16:1 supplement (Experimental): Volunteers will take cis-C16:1 supplement for 3 weeks
  Interventions: Dietary Supplement: Cis-C16:1 supplement

INTERVENTIONS:
Dietary Supplement: Trans-C16:1 supplement — Each volunteer will consume 3 escalating doses (120 mg/day, 240 mg/day and 480 mg/day) of trans-C16:1 enriched vegetable oil for 3 weeks each (3 doses x 3 weeks each [9 weeks total]
  Arms: Trans-C16:1 supplement
Dietary Supplement: Cis-C16:1 supplement — Each volunteer will consume 3 escalating doses (380 mg/day, 760 mg/day and 1520 mg/day) of cis-C16:1 enriched vegetable oil for 3 weeks each (3 doses x 3 weeks each [9 weeks total]
  Arms: Cis-C16:1 supplement

SUMMARY:
Trans-palmitoleic acid (trans-C16:1) is a naturally occurring trans fatty acid present in small quantities in foods, most notably in dairy products. Observational evidence suggests a positive association between trans-C16:1 and insulin sensitivity, and negative association with risk of developing type 2 diabetes mellitus [1-3]. Cis-palmitoleic acid (cis-C16:1) is found naturally in foods and is particularly high in macadamia nuts and oil extracted from the sea buckthorn plant. Animal models suggest that this palmitoleic acid isomer also improves insulin sensitivity and reduces metabolic dysfunction.

This pilot dosing study is necessary to inform the design of a larger trial to test the hypothesis that both trans-C16:1 and cis-C16:1 improve insulin resistance but at different doses. Plasma phospholipid fatty acid profiles will be used as the primary outcome measure.

DETAILED DESCRIPTION:
The fatty acids trans-C16:1 and cis-C16:1 have been associated with healthy plasma glucose levels. Elevated glucose levels have been associated with diabetes. This study is designed to determine whether there is a dose-response relation between how much trans-C16:1 and cis-C16:1 you consume and how much appears in plasma. This information will be used to design a future study to determine whether trans-C16:1 and cis-C16:1 could be used to treat diabetes. Trans-C16:1 occurs naturally in dairy fat such as milk and cheese, while cis-C16:1 occurs naturally in nuts, particularly, macadamia nuts, and a plant called sea buckthorn. The study will consist of two 9-week phases, with a minimum of a 4 week off-study period between the two phases. Fasting blood will be drawn at baseline (first day of week 1), 3 weeks, 6 weeks and 9 weeks (4 total blood draws per phase or 8 total blood draws for 2 phases). During each phase you will be asked to consume increasing numbers of vegetable oil capsules, 2 per day during the first 3 weeks, 4 per day during the second 3 weeks, and 8 per day during the third 3 weeks. During each of these periods you should take half the capsules in the morning and half in the evening, with your meals. You will be randomly assigned to receive the trans-C16:1 or cis-C16:1 during the first phase and the other during the second phase. The total length of the study is about 18 weeks, not including the break between phase 1 and phase 2 (not less than 4 weeks). The trans-C16:1 in the capsules will be in the form of partially-hydrogenated soybean oil. The cis-C16:1 in the other capsules will be in the form of sea buckthorn oil.

ELIGIBILITY:
1. Inclusion criteria:

   * Age ≥ 18 to ≤ 70 years
   * BMI ≥ 25 kg/m2 ≤ 40 kg/m2
   * Normotensive with or without medication
   * Normal fasting plasma glucose levels (≤120 mg/dL)
   * Normal kidney function as assessed by serum creatinine and blood urea nitrogen
   * Normal liver function as assessed by serum glutamic pyruvic transaminase (SGPT), serum glutamic oxaloacetic transaminase (SGOT) and alkaline phosphatase (ALP)
   * Normal thyroid function defined as screening TSH within normal ranges, without or with medication for at least 6 months
   * Normal gastrointestinal function
2. Exclusion criteria:

   * Use of supplements containing fish oil or other lipid supplements (e.g., flaxseed, primrose oil, sea buckthorn oil) within 3 months of study participation
   * Greater than 2 servings/day combined of cheese, whole-fat milk or whole-fat yogurt
   * Diagnosed diabetes mellitus Type I or Type II and/or taking glucose lowering medications (e.g., metformin, actos, januvia)
   * Use of medication known to affect lipid metabolism (HMG-CoA reductase inhibitors (statins, red yeast rice), bile acid sequestrants, cholesterol absorption inhibitors (exetimibe [Zetia]), nicotinic acid agents, fibrates, probucol, anticoagulants, hormone therapy medications containing estrogen, anabolic steroids)
   * Established major chronic diseases such as major cardiovascular disease (history of myocardial infarction, stroke, symptomatic heart failure, coronary artery bypass graft, or symptomatic peripheral arterial disease), active cancer, end stage renal disease, dementia, severe chronic obstructive pulmonary disease, significant liver disease
   * Pregnancy or breastfeeding
   * Unwillingness to adhere to study protocol
   * No Social Security number (for payment and IRS forms).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2015-07; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Plasma phospholipid fatty acid profiles - | 18 weeks
  PLP FA profile determined by gas chromatography

SECONDARY OUTCOMES:
Plasma sphingolipid profiles - | 18 weeks
  sphingolipid profile determined by qTOF (quadrupole time of flight mass spectrometry)
CBC | 18 weeks
  complete blood count
Insulin | 18 weeks
  determined by ELISA
Clinical Chemistry Profile | 18 weeks
  glucose, albumin, ALP, SGPT, SGOT, blood urea nitrogen, creatine phosphokinase, creatinine, lactate dehydrogenase, total protein, bilirubin, globulin, albumin/globulin ratio, uric acid, calcium, phosphorus, magnesium, sodium, potassium, chloride, total and LDL-cholesterol, triglyceride
HDL-cholesterol | 18 weeks
  automated immunoturbidimetric assay
glucose | 18 weeks
  part of chemistry panel
albumin | 18 weeks
  part of chemistry panel
ALP | 18 weeks
  alkaline phosphatase - part of chemistry panel
SGPT | 18 weeks
  serum glutamic pyruvic transaminase - part of chemistry panel
SGOT | 18 weeks
  serum glutamic oxaloacetic transaminase - part of chemistry panel
blood urea nitrogen | 18 weeks
  assessment of kidney function - part of chemistry panel
creatine phosphokinase | 18 weeks
  muscle enzymes - part of chemistry panel

CONTACTS AND LOCATIONS:
Overall Officials: Alice H Lichtenstein, D.Sc., Principal Investigator — Tufts University/Jean Mayer Human Nutrition Research Center on Aging
Locations (1):
- Jean Mayer Human Nutrition Research Center on Aging, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huang NK, Matthan NR, Galluccio JM, Shi P, Lichtenstein AH, Mozaffarian D. Supplementation with Seabuckthorn Oil Augmented in 16:1n-7t Increases Serum Trans-Palmitoleic Acid in Metabolically Healthy Adults: A Randomized Crossover Dose-Escalation Study. J Nutr. 2020 Jun 1;150(6):1388-1396. doi: 10.1093/jn/nxaa060. PMID 32140719